CLINICAL TRIAL: NCT04576208
Title: A Randomized Open-label Phase 2 Multicenter Study to Evaluate the Impact of Management Strategies on Gastrointestinal-Related Adverse Events in Patients With Non-Small Cell Lung Cancer Harboring EGFR Exon 20 Insertion Mutations Receiving TAK-788
Brief Title: A Study to Evaluate the Impact of Management Strategies on Gastrointestinal-Related Adverse Events in Participants With Non-Small Cell Lung Cancer Harboring Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertion Mutations Receiving TAK-788
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision (no safety or efficacy concerns)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TAK-788-2001; 2020-002045-41 (EudraCT Number); U1111-1251-7658 (Other: WHO)
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — mobocertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): TAK-788 160 mg, capsules, orally, once daily (QD) with or without a low-fat meal until disease progression or as assessed by the investigator during every 3-week cycle.
  Interventions: Drug: TAK-788
- Cohort 2 (Experimental): TAK-788 160 mg, capsules, orally, QD with or without a low-fat meal and antidiarrheal prophylaxis administered during the first 8 weeks of treatment until disease progression or as assessed by the investigator during every 3-week cycle.
  Interventions: Drug: TAK-788; Drug: Antidiarrheal prophylaxis

INTERVENTIONS:
Drug: TAK-788 — TAK-788 capsules
  Other Names: AP32788; Mobocertinib
Drug: Antidiarrheal prophylaxis — Antidiarrheal prophylaxis includes loperamide tablet administered as per routine clinical practice.
  Arms: Cohort 2

SUMMARY:
The purpose of the study is to characterize the incidence and severity of TAK-788-associated diarrhea in previously treated participants with locally advanced or metastatic non-small-cell lung cancer (NSCLC) whose tumors harbor EGFR exon 20 insertion mutations treated with TAK-788 when administered with or without intensive loperamide prophylaxis.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-788. TAK-788 administered with or without antidiarrheal prophylaxis is being tested to evaluate the impact of management strategies on gastrointestinal-related adverse events in participants with non-small cell lung cancer harboring EGFR Exon 20 insertion mutations receiving TAK-788.

The study will enroll approximately 90 patients. Participants will be randomly assigned in 1:1 ratio (by chance, like flipping a coin) to one of the two treatment groups-

* Cohort 1
* Cohort 2

All participants will be asked to take TAK-788 capsules with or without a low-fat meal in Cohort 1 and TAK-788 capsule with antidiarrheal prophylaxis and with or without a low-fat meal in Cohort 2.

This is a multi-center trial and will be conducted worldwide. The overall time to participate in this study is approximately 2 years. Participants will make multiple visits to the clinic after receiving their last dose of drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with histologically or cytologically confirmed nonsquamous cell locally advanced (not suitable for definitive therapy) or metastatic non-small-cell lung cancer (NSCLC) (Stage IIIB or IV) NSCLC; and, has received at least 1 prior line of therapy for this disease.
2. A documented epidermal growth factor receptor (EGFR) mutation with in-frame exon 20 insertion, confirmed as follows:

   * For sites located in the United States (US): assessment must be done by a certified laboratory functioning under the guidelines of the Clinical Laboratory Improvements Amendment (CLIA).
   * For site located outside of the US: assessment must be done by an accredited local laboratory.

   Note: A documented EGFR in-frame exon 20 insertion or insertion-duplication includes but is not limited to one of the following:
   * A763_Y764insFQEA,
   * V769_D770insASV (also referred to as ASV duplication)
   * D770_N771insNPG
   * D770_N771insSVD (also referred to as SVD duplication)
   * H773_V774insNPH (also referred to as NPH duplication), or
   * Any other in-frame insertion mutation in the exon 20 [amino acids 739 -823].

   The EGFR exon 20 insertion mutation can be either alone or in combination with other EGFR or HER2 mutations. The reported insertion-duplication can have been detected on either tissue or liquid biopsy using a well-validated test based on either polymerase chain reaction, sequencing or next-generation sequencing (NGS).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Minimum life expectancy of ≥3 months.
5. All toxicities from prior therapy have been resolved to ≤Grade 1, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 or have resolved to baseline, at the time of first dose of TAK-788.

Exclusion Criteria:

1. Has been diagnosed with another primary malignancy other than NSCLC, except for the following:

   1. Adequately treated non-melanoma skin cancer or cervical cancer in situ.
   2. Definitively treated non-metastatic prostate cancer.
   3. Non-NSCLC primary malignancies that are definitively relapse-free for ≥3 years.
2. Has unstable brain metastases to include previously untreated intracranial central nervous system (CNS) metastases or previously treated intracranial CNS metastases with radiologically documented new or progressing CNS lesions.

   - Brain metastases that are stable do not preclude eligibility if they have been treated with surgery and/or radiation, and have been stable without requiring corticosteroids to control symptoms within 7 days before randomization, and have no evidence of new or enlarging brain metastases.
3. Has a current spinal cord compression (symptomatic or asymptomatic that is detectable by radiographic imaging) or leptomeningeal disease (symptomatic or asymptomatic).
4. Currently has or has had a history of interstitial lung disease, to include radiation or drug related pneumonitis that requires/required steroid treatment.
5. Has an ongoing or active infection, to include but not limited to infections requiring intravenous antibiotics or has a known history of HIV. Testing for HIV is not required in the absence of history.

   Note: Hepatitis B surface antigen-positive participants are allowed to enroll if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is below 1000 copies/mL in the plasma. Patients who are positive for anti-hepatitis C virus antibody can be enrolled but must not have detectable hepatitis C virus (HCV) RNA in the plasma.
6. Have uncontrolled hypertension. Participants with hypertension should be under treatment on study entry to control blood pressure.
7. A prolonged QTcF interval, or is being treated with medications known to be associated with the development of Torsades de Pointes.
8. Has a GI illness or disorder, including but not limited to a history of GI perforation, that could affect oral absorption of TAK-788.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) of ≥Grade 3 Diarrhea Occurring During the First 4 Cycles of TAK-788 Dosing | Approximately 15 Months
  An Adverse Event (AE) is defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Grading will be done using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria. Per NCI CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.

SECONDARY OUTCOMES:
Number of Participants with TEAEs of ≥Grade 3 Nausea and Vomiting Occurring During the First 4 Cycles of TAK-788 Dosing | Approximately 15 Months
  An AE is defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Grading will be done using the NCI-CTCAE criteria. Per NCI CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Number of Participants With TEAEs of Diarrhea, Nausea, Vomiting and Other Adverse Event of Clinical Interest (AECIs) Occurring During the First 4 Cycles of TAK-788 Dosing | Approximately 15 Months
  An AE is defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Overall Response Rate (ORR) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Approximately 15 Months
  ORR will be defined as the percentage of participants achieving complete response (CR) or partial response (PR). CR is defined as disappearance of all extranodal target lesions. PR is defined as at least a 30% decrease in Sum of the Longest Diameters (SLD) of target lesions, taking as a reference the baseline SLD.
Duration of Response as per RECIST Version 1.1 | Approximately 15 Months
  DOR will be defined as the time interval from the time that the measurement criteria are first met for CR or PR (whichever is first recorded) until the first date that PD is objectively documented. CR is defined as disappearance of all extranodal target lesions. PR is defined at least a 30% decrease in Sum of the Longest Diameters (SLD) of target lesions, taking as a reference the baseline SLD. PD is defined as at least a 20% increase in the Sum of Diameters (SoD) of target lesions, taking as a reference the smallest (nadir) SoD since (and including) baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm.
Progression Free Survival (PFS) as per RECIST Version 1.1 | Approximately 15 Months
  PFS will be defined as the interval from the randomization date until the first date at which the criteria for disease progression according to RECIST version 1.1 are met or death. PD is defined as at least a 20% increase in the SoD of target lesions, taking as a reference the smallest (nadir) SoD since (and including) baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm.
Health-Related Quality of Life (HRQoL) as Assessed European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 Score | Approximately 15 Months
  The EORTC QLQ-C30 is a cancer-specific questionnaire tested in participants with lung cancer. The EORTC QLQ-C30 will be scored for 5 functional scales (physical, role, cognitive, emotional, and social functioning); 3 symptom scales (fatigue, pain, and nausea/vomiting); and a global health status/quality-of-life (QoL) scale. Six single-item scales are also included (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Raw scores are converted into scale scores ranging from 0 to 100. For the functional scales and the global health status/QoL scale, higher scores represent better HRQoL, whereas for the symptom scales lower scores represent better HRQoL.
Health-Related Quality of Life (HRQoL) as Assessed by EORTC Lung Cancer Module (QLQ-LC13) Score | Approximately 15 Months
  The EORTC QLQ-LC13 module will comprise 13 questions assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and use of pain medication. The LC13 module incorporates 1 multi-item scale to assess dyspnea, and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and haemoptysis. Raw scores are converted into scale scores ranging from 0 to 100, where the higher scores represent worse symptoms and lower scores represent better HRQoL.
Health-Related Quality of Life (HRQoL) as Assessed by Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) Score | Approximately 15 Months
  The NSCLC-SAQ is qualified by the US Food and Drug Administration (FDA) to measure symptoms of NSCLC. The NSCLC-SAQ has 7 items with 5-level verbal rating scale and measures the severity/frequency of the following NSCLC symptoms: cough, pain, dyspnea, fatigue, and appetite. The raw scores are ranged from 0 to 4 and total score is ranged from 0-20.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/